CLINICAL TRIAL: NCT06405880
Title: Implementation of Pharmacist Case Finding and Intervention for Vascular Prevention (PRxOACT) Study
Brief Title: Pharmacist Case Finding and Intervention for Vascular Prevention Trial
Acronym: PRxOACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00139142
Record Dates: First submitted 2024-05-01; First posted 2024-05-09 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Risk Factors; Blood Pressure; Cardiovascular Disease; Diabetes; Dyslipidemia
Keywords: cardiovascular; blood pressure; diabetes; dyslipidemia
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Dyslipidemias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist-led care pathway (Experimental): Participants in the intervention arm will receive the care using a shared decision-making pharmacist-led care pathway designed to guide the cardiovascular (CV) risk reduction process. The pharmacist-led care pathway is modelled after the largest CV risk reduction randomized controlled trial in a community pharmacy setting (RxEACH Study), and based upon the latest CV risk reduction guidelines, such as C-CHANGE. This pathway will be built into a computer web-based program and include step-by-step, algorithm-guided patient assessment to calculate the participant's estimated CV risk. The participant and pharmacist will be guided by the care pathway to review the participant's estimated CV risk and contributing CV risk factors and engage in shared decision-making to manage the participant's CV risk factors using lifestyle changes and/or pharmacological treatment as clinically appropriate.
  Interventions: Other: Pharmacist-led care pathway
- Usual Care (No Intervention): The control group will involve facilitated relay of information to participants' family physician. Participants in the control group will have their pharmacist collect information informing the patient's CV risk. Participants will then be given a letter that contains their values for CV risk factors (including blood pressure, HbA1c, and lipid panel), and they will be advised to present it to their family physician. No specific suggestions for CV risk reduction will be detailed in the letter. In the case where the patient does not have a family physician, they can be referred to a physician walk-in clinic. A follow-up appointment in 6-months' time will be booked for with all participants in the control group.

INTERVENTIONS:
Other: Pharmacist-led care pathway — Participants in the intervention arm will receive the care using a shared decision-making pharmacist-led care pathway designed to guide the cardiovascular (CV) risk reduction process. The pharmacist-led care pathway is modelled after the largest CV risk reduction randomized controlled trial in a community pharmacy setting (RxEACH Study), and based upon the latest CV risk reduction guidelines, such as C-CHANGE. This pathway will be built into a computer web-based program and include step-by-step, algorithm-guided patient assessment to calculate the participant's estimated CV risk. The participant and pharmacist will be guided by the care pathway to review the participant's estimated CV risk and contributing CV risk factors and engage in shared decision-making to manage the participant's CV risk factors using lifestyle changes and/or pharmacological treatment as clinically appropriate.
  Arms: Pharmacist-led care pathway

SUMMARY:
Heart disease is a common and serious medical condition which causes nearly one in every three deaths worldwide every year.

The factors which increase people's risk for heart disease are well-known, but there needs to be more support given to people to reduce their risk of heart disease. Pharmacists are front line primary healthcare providers who see patients more frequently than any other healthcare provider and can help people reduce their risk of heart disease.

This research project aims to see whether a pharmacist-led intervention can help people reduce their risk of heart disease. The potential impact of this project is to empower people to understand how to reduce their risk of heart disease and reduce the burden of heart disease on the community.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older)
* Clinical diagnosis of at least one of the following conditions:

  * Diabetes,
  * Chronic kidney disease,
  * Chronic inflammatory condition (e.g., rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, gout, systemic lupus erythematosus or psoriasis),
  * Atherosclerotic vascular disease,
  * Hypertension,
  * Obesity (defined as body mass index greater than 30),
  * Current tobacco or vape use

Exclusion Criteria:

* Unwilling to participate/sign consent form;
* Unwilling or unable to participate in regular follow-up visits; or
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1003 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Estimated cardiovascular risk | Up to 6 months.
  The primary outcome is the difference in change in estimated CV risk (calculated using the EPI·RxISK™ calculator: https://www.epicore.ualberta.ca/epirxisk/) from baseline to the end of the study (up to six months) between the intervention and control groups.

SECONDARY OUTCOMES:
A1c in those who have diabetes | Up to 6 months.
  The difference in change in serum A1c in those who have diabetes from baseline to the end of the study (up to six months) between the intervention and control groups
Blood pressure | Up to 6 months.
  The difference in change in blood pressure from baseline to the end of the study (up to six months) between the intervention and control groups
LDL Cholesterol Concentration | Up to 6 months.
  The difference in change in serum LDL-cholesterol concentration from baseline to the end of the study (up to six months) between the intervention and control groups
Tobacco use or vaping | Up to 6 months.
  The difference in the proportion of participants who report tobacco or vape use from baseline to the end of the study (up to six months) between the intervention and control groups.
Yield of enrolment approaches | Up to 6 months.
  The yield from each enrolment approach used (active case-finding approach vs. passive approaches such as when the patient attends the pharmacy to collect a prescription medication or through patient self-identification)
Yield of enrollment by pharmacy type | Up to 6 months.
  Yield of enrollment by clinic or non-clinic pharmacy type
Shared-decision making uptake | Up to 6 months.
  Extent to which shared decision making was achieved in the intervention as measured by the validated Shared Decision Making 9-item Questionnaire (SDM-Q-9) tool. The minimum score is 0 and the maximum score is 45, where a higher score indicates a greater subjective level of shared decision making.
Previous cardiovascular risk assessment | Up to 6 months.
  Proportion of participants who never had their cardiovascular risk assessed before the study.
Proportion categorized as having high cardiovascular risk | Up to 6 months.
  Proportion of participants who are categorized as having high cardiovascular risk.
Patient satisfaction | Up to 6 months.
  Patient satisfaction as measured by the Consultation Satisfaction Questionnaire. Minimum score is 18 and maximum score is 90, where a higher score indicates higher patient satisfaction.
Types of intervention delivered by the pharmacist | Up to 6 months.
  Types of interventions provided by the pharmacists, such as education on lifestyle factors (tobacco cessation, diet, exercise), prescribing or changing the dose of medications, education on new or changed medications, education on adherence to medications and/or lifestyle recommendations.
Quality of life reported by study participants | Up to 6 months.
  The difference in change in quality of life as measured using the validated EuroQoL 5 Dimensions 5 Levels (EQ-5D-5L) Scale between the intervention and control groups. The EQ-5D-5L will be scored by collecting individuals' health state index value, which will be converted into an EQ 5D summary value according to the preferences of the general population of a country/region.

CONTACTS AND LOCATIONS:
Overall Officials: Ross Tsuyuki, Study Director — University of Alberta; Yazid Al Hamarneh, Principal Investigator — University of Alberta
Locations (1):
- The University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Liu S, Tsuyuki RT, Graham MM, Nelson D, Semeniuk G, Al Hamarneh YN. Implementation of Pharmacist Case-Finding and Care Pathway Intervention for Vascular Prevention (PRxOACT): Protocol for a Randomized Controlled Trial. CJC Open. 2025 Mar 20;7(6):821-831. doi: 10.1016/j.cjco.2025.03.011. eCollection 2025 Jun. PMID 40586019